CLINICAL TRIAL: NCT00602706
Title: A Phase I/II Dose Escalation Study Assessing the Toxicity and Efficacy of 153-Samarium-EDTMP in Place of TBI in the Conditioning Regimen for PBSCT for Patients With Multiple Myeloma
Brief Title: Samarium Sm 153 Lexidronam Pentasodium and High-Dose Melphalan in Treating Patients With Multiple Myeloma Undergoing Stem Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Angela Dispenzieri, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000582552; P30CA015083 (NIH); MC9981 (Other: Mayo Clinic Cancer Center); 1046-99 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — sargramostim; Melphalan; Peripheral Blood Stem Cell Transplantation; samarium Sm-153 lexidronam

INTERVENTIONS:
Biological: sargramostim
Drug: melphalan
Procedure: autologous hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: samarium Sm 153 lexidronam pentasodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells either by killing the cells or by stopping them from dividing. Samarium Sm 153 lexidronam pentasodium contains a radioactive substance that kill cancer cells. Peripheral blood stem cell transplant using stem cells from the patient may be able to replace immune cells that were destroyed by chemotherapy and radioactive drugs used to kill cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of samarium Sm 153 lexidronam pentasodium when given together with high-dose melphalan in treating patients with multiple myeloma undergoing stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To find the maximum tolerated dose of samarium Sm 153 lexidronam pentasodium when given with fixed high-dose melphalan as a conditioning regimen for autologous peripheral blood stem cell transplantation in patients with multiple myeloma. (Phase I)
* To assess the response rates of this regimen in these patients. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of samarium Sm 153 lexidronam pentasodium followed by a phase II study.

* Phase I: Patients receive samarium Sm 153 lexidronam pentasodium IV once between days -14 and -10. Patients also receive melphalan IV on day -1. Patients undergo peripheral blood stem cell transplantation on day 0. Patients receive sargramostim (GM-CSF) subcutaneously once daily beginning on day 6 and continuing until blood counts recover.
* Phase II: Patients receive samarium Sm 153 lexidronam pentasodium at the MTD determined in phase I .

Blood samples are collected periodically to determine clearance of samarium Sm 153 lexidronam pentasodium and bone marrow dosimetry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma requiring treatment
* Must have at least 2 x 10^6 CD34+ cells collected for peripheral blood stem cell transplantation

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-2 (ECOG PS > 2 allowed if secondary to neuropathy or acute bone event)
* Direct bilirubin ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 750 μ/L
* Creatinine ≤ 3.0 mg/dL
* Ejection fraction ≥ 45%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 6 months after the completion of study therapy

Exclusion criteria:

* DLCO < 50%
* FVC < 50%
* FEV_1 < 50%
* Active malignancy with the exception of nonmelanoma skin cancer
* Uncontrolled infection
* NYHA class III-IV cardiac disease

PRIOR CONCURRENT THERAPY:

* May or may not have received prior chemotherapy
* At least 3 weeks since prior chemotherapy

  * Cyclophosphamide pulsing for stem cell collection allowed
* At least 4 weeks since prior biologic therapy
* At least 2 weeks since prior bisphosphonates and bisphosphonates maybe resumed 1 month post-study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2000-01; Primary Completion 2003-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of toxicity incidents (Phase I)
Proportion of successes (Phase II)

SECONDARY OUTCOMES:
Number of responses (Phase I)
Overall survival (Phase II)
Progression-free survival (Phase II)
Time to progression (Phase II)
Progressive disease variables

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, MD, Study Chair — Mayo Clinic